CLINICAL TRIAL: NCT02837458
Title: Application of High Frequency Electrical Currents: Effects on Mechanical Threshold, Tactile Threshold and Evoked Potentials in Healthy Subjects.
Brief Title: Effect of High Frequency Electrical Currents in Healthy Subjects.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Castilla-La Mancha (Other)
Collaborators: Hospital Nacional de Parapléjicos de Toledo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ddsm18
Record Dates: First submitted 2016-07-15; First posted 2016-07-19 (Estimated); Last update posted 2020-02-19 (Actual); Status verified 2017-04

CONDITIONS: High Frequency Current
Keywords: Electric current; Nerve block; somatosensory evaluation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-Frequency (Experimental): Transcutaneous application of high frequency electrical current over the arm for a 30 minutes session. The intensity of the current will increase until participants report a "strong but comfortable" sensation, just below motor threshold.
  Interventions: Device: High-Frequency
- Sham Stimulation (Sham Comparator): Electrodes are placed over the arm for a 30 minutes in the same manner as experimental group but will be applied a sham electrical stimulation increasing the current intensity of an unconnected channel.
  Interventions: Device: Sham Stimulation

INTERVENTIONS:
Device: High-Frequency — high-Frequency electrical stimulation over superficial radial nerve through the electrotherapy device Myomed 932. (Enraf-Nonius, Delft, Netherlands)
  Arms: High-Frequency
Device: Sham Stimulation — Sham transcutaneous electrical stimulation over superficial radial nerve through the electrotherapy device Myomed 932. (Enraf-Nonius, Delft, Netherlands)
  Arms: Sham Stimulation

SUMMARY:
The purpose of this study is to determine whether the transcutaneous application of unmodulated high frequency alternating currents could produce a quickly conduction block of peripheral nerve.

DETAILED DESCRIPTION:
In the last years several animal experimental studies have evidenced that high frequency unmodulated currents about 5 KHz can cause a peripheral nerve block. However electric currents with these high frequencies that are usually used for the treatment of pain in humans are interrupted or modulated (i.e. interferential currents).

It has show that the diameter of the nerve it is related with the frequency to produce the conduction block. For this reason we decided to applied 30KHz to observe the effects on pain in patients with whiplash and to compare versus sham stimulation.

Only one study has applied 5KHz on experimental pain and they have demonstrated changes in somatosensory thresholds.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

Exclusion Criteria:

* Neuromuscular disease.
* Epilepsy.
* Trauma, surgery or pain affecting the upper limb, shoulder girdle or cervical area.
* Osteosynthesis material in the upper limb.
* Diabetes.
* Cancer.
* Cardiovascular disease.
* Pacemaker or other implanted electrical device.
* Take any drug (NSAIDs, corticosteroids, antidepressants, analgesics, antiepileptics, ...) during the study and in the previous 7 days.
* Presence of tattoos or other external agent introduced into the treatment or assessment area.
* Pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
Baseline Mechanical Pain Threshold | baseline at 0 min
  The pressure pain threshold will be measured by a pressure algometer and will be expressed in Newton
Baseline Tactile Threshold | baseline at 0 min
  The tactile threshold will be measured with Von Frey filaments and will be expressed in millinewton
Baseline Muscle Strength | Baseline at 0 min
  The muscle strength will be measured with a dynamometer and will be expressed in Newton
Mechanical Pain Threshold after treatment at 30 min | Immediately after treatment at 30 min
  The pressure pain threshold will be measured by a pressure algometer and will be expressed in Newton
Tactile Threshold after treatment at 30 min | Immediately after treatment at 30 min
  The tactile threshold will be measured with Von Frey filaments and will be expressed in millinewton
Muscle Strength after treatment at 30 min | Immediately after treatment at 30 min
  The muscle strength will be measured with a dynamometer and will be expressed in Newton

SECONDARY OUTCOMES:
Change from baseline in Mechanical Pain Threshold | baseline at 0 min, immediately after treatment at 30 min
  The pressure pain threshold will be measured by a pressure algometer and will be expressed in Newton
Change from baseline in TactileThreshold | baseline at 0 min, immediately after treatment at 30 min
  The tactile threshold will be measured with Von Frey filaments and will be expressed in millinewton
Change from baseline in Muscle strength | baseline at 0 min, immediately after treatment at 30 min
  The muscle strength will be measured with a dynamometer and will be expressed in Newton

CONTACTS AND LOCATIONS:
Overall Officials: Diego Serrano-Muñoz, MsC, Principal Investigator — Hospital Nacional de Parapléjicos, Toledo
Locations (1):
- Diego Serrano-Muñoz, Toledo, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Serrano-Munoz D, Avendano-Coy J, Simon-Martinez C, Taylor J, Gomez-Soriano J. 20-kHz alternating current stimulation: effects on motor and somatosensory thresholds. J Neuroeng Rehabil. 2020 Feb 19;17(1):22. doi: 10.1186/s12984-020-00661-x. PMID 32075666